CLINICAL TRIAL: NCT01890460
Title: Quantitative Evaluation of Liver Disease With Liver Elastography Measurements Using the Supersonic Imagine Aixplorer ShearWaveTM Elastography Ultrasound Machine in Patients Undergoing Liver Transplant Surgery
Brief Title: Evaluation of Liver Disease With Elastography Measurements in Patients Undergoing Liver Transplant Surgery
Acronym: SupersonicOR
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 013-041
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to compare ultrasound measurements of the liver obtained prior to surgery on the skin to measurements obtained during surgery directly on the diseased liver. The objective is to determine if ultrasounds of the liver on the skin can provide accurate measurements of disease of the liver to provide an alternative option to liver biopsies.

DETAILED DESCRIPTION:
A non-invasive, ultrasound platform based, ShearWaveTM Elastography measurement will be obtained at two time points on each qualified patient. The first time point will be in the operating room before the initial incision is made. The second time point involves placement of a small, hand-held modified ultrasound probe directly on the patient's diseased liver during the liver transplant surgery. The probe used in this study is the SuperCurved™SC6-1, capable of a band width of 1-6MHz with 192 elements.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18
* Patients undergoing a liver transplant surgery

Exclusion Criteria:

* Any person unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a liver transplant surgery
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To obtain quantitative evaluation of the progression of liver disease, using ShearWaveTM Elastography measurements obtained with the Supersonic Imagine Aixplorer ultrasound machine in patients undergoing a liver transplant surgery. | on day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: James Trotter, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided